CLINICAL TRIAL: NCT02586870
Title: Assessment of Renal Artery Fibromuscular Dysplasia: From Diagnosis to Treatment
Acronym: DysArt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-A01244-45; 2015-14 (Other: assistance publique hopitaux de marseille)
Record Dates: First submitted 2015-10-22; First posted 2015-10-27 (Estimated); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Renal Artery Fibromuscular Dysplasia
MeSH Terms: interventions — Ultrasonography, Interventional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Intravascular Ultrasound

SUMMARY:
This is a prospective multicenter study based on the validation of diagnostic criteria and predictive factors of treatment efficacy for renal artery stenosis in renal artery dysplasia. This is considered as a rare disease and patients are usually treated in specialized centers involved in a national network. Marseille is a center specialized in FMD and a member of the network that is very active across the country. In order to rapidly recruit patients the investigators propose a multicenter study. All patients included will benefit from an invasive angiography with trans stenotic gradient assessment at rest. In case of bilateral stenosis the investigators will randomly omit data from one side and consider the data from the contralateral artery for further analysis, to avoid statistical interdependency. Patients who require angioplasty and who have unilateral stenosis (unilateral FMD lesion or bilateral but with one non significant stenosis based on duplex ultrasound European recommendations for atherosclerotic renal artery stenosis) will be included in the second part of the study. These patients will in addition benefit from a trans stenotic pressure assessment under vasodilation and intravascular renal artery ultrasound. Patients with severe bilateral renal artery stenosis will not be included in the analysis to assess predictive criteria for treatment efficacy on hypertension, treatment of these patients will followed the current best clinical practice. These patients will be followed during 6 to 8 month to assess potential complication of the pressure assessment renal artery stenosis, but their data will be included to assess the value of FFR and IVUS to guide the procedure. Patients with unilateral stenosis will be followed up 6 month after angioplasty in order to assess hypertension and to look for potential complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* hypertension based on ambulatory BP 24H measurements (12h mean daytime BP ≥135 or 85 mmHg)
* renal artery stenosis due to multifocal FMD of the main renal artery or accessory artery with a diameter ≥ 5mm (defined using CT scan or duplex ultrasound),
* if clinical and para-clinical information suggest that the hypertension might be caused by the renal stenosis and will require intravascular revascularization because of:
* Recent onset of hypertension
* Resistant hypertension (hypertension treated by 3 hypertensive drugs including one diuretic) based on ambulatory BP measurements (12h mean daytime BP ≥135 or 85 mmHg)
* Hypertension for patients with poor compliance to medications or medication side effects.
* Acute flash pulmonary edema
* Delayed onset of hypertension with a decrease in kidney size or recent onset of renal failure especially after a renin-angiotensin system blocker

Exclusion Criteria:

* Patients with other causes of secondary hypertension
* Patients with renal artery stenosis from other causes than FMD higher than 30%
* Patients with unifocal FMD or intimal FMD
* Multifocal FMD of an accessory renal artery with a diameter < than 5 mm.
* Patient with involvement of a collateral artery of the main renal artery
* Renal artery dissection
* Patients with creatinine clearance (MDRD) lower that 40ml/min/1.73m2.
* Patients with an aneurysm with a diameter more than twice the diameter of the concerned artery
* Patients without a social security number
* Pregnant patients
* Patients who refuse to participate in the study
* Patients for whom the invasive measure are not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-11; Primary Completion 2020-02-02 (Actual); Study Completion 2020-02-02 (Actual)

PRIMARY OUTCOMES:
MAXIMAL VELOCITY | 24 months
  duplex ultrasound parameters
ratio between maximal speed in the renal artery and in the aorta | 24 MONTHS
  duplex ultrasound parameters
resistance index | 24 MONTHS
  duplex ultrasound parameters
systolic ascension time | 24 MONTHS
  duplex ultrasound parameters

SECONDARY OUTCOMES:
stenosis length | 24 months
  MDCT anatomical parameters
arterial diameter | 24 MONTHS
  MDCT anatomical parameters
number of the stenosis | 24MONTHS
  MDCT anatomical parameters
Distance Ostium / main stenosis | 24 MONTHS
  MDCT anatomical parameters

CONTACTS AND LOCATIONS:
Overall Officials: catherine GEINDRE, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Cadour F, Silhol F, Iline N, Giorgi R, Lorthioir A, Amar L, Sapoval M, Rousseau H, Sarlon G, Thony F, Jacquier A. Insights from intravascular pressure measurement of renal artery revascularization in patients with fibromuscular dysplasia: The DYSART study. J Vasc Surg. 2022 Mar;75(3):939-949.e1. doi: 10.1016/j.jvs.2021.09.023. Epub 2021 Sep 30. PMID 34601043